CLINICAL TRIAL: NCT02186197
Title: The Impact of Fellow-performed Cardiopulmonary Ultrasound Exams on the Diagnosis and Management of Shock and Respiratory Failure
Brief Title: The Impact of Fellow-performed Cardiopulmonary Ultrasound Exams
Status: Completed | Type: Observational
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 206-13
Record Dates: First submitted 2014-06-25; First posted 2014-07-10 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Shock; Respiratory Failure
Keywords: Volume Responsiveness
MeSH Terms: conditions — Shock; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Shock and/or Respiratory Failure
  Interventions: Other: Critical Care Ultrasound

INTERVENTIONS:
Other: Critical Care Ultrasound — A critical care ultrasound exam will be performed on all patients included in this study

SUMMARY:
Shock and respiratory failure are common reasons for admission to the intensive care unit (ICU) at our institution. The various causes of acute shock and respiratory failure are traditionally assessed with the use of history, physical examination, chest x-ray, EKG and laboratory studies. Unfortunately, much of this clinical information is either insensitive or non-specific. 1 Critical care ultrasound (CCUS) is a rapid and non-invasive tool, which has been shown to be useful in the intensive care unit to assist in the diagnosis and management of patients in shock or respiratory failure.2

The investigators hypothesize that the trained fellow's interpretation of critical care ultrasound images will be accurate when compared to experts and that ultrasounds will change diagnosis and management of the patient in shock and respiratory failure.

DETAILED DESCRIPTION:
In recent years, CCUS has become widely used by clinicians in the field of critical care as a rapid and non-invasive tool for providing diagnostic information. At Beth Israel Medical Center, CCUS has been routinely used for over a decade on a daily basis by both fellows and attending to aid in the diagnosis and management of shock and respiratory failure.

Numerous studies have described the accuracy and speed of clinician-performed critical care ultrasound. Recently it was shown that early critical care ultrasound by attendings can modify admitting diagnosis and in many cases change management. This study was done by expert practitioners and not by trainees. The accuracy of fellow image interpretation or the proportion of time that a fellow-performed ultrasound exam changes diagnosis or management has not been studied.

The protocol used in this study has already been implemented as part of the diagnostic assessment of a critically ill patients in our care and as an educational tool to help fellows learn ultrasound. The goal of this study is organize the existing clinical data to determine the accuracy of fellow interpretation along with the diagnostic impact of fellow performed CCUS.

Methods:

This is an observational study to see how accurately subjects (fellows) perform CCUS and what impact CCUS has on the early diagnosis of shock and respiratory failure in our ICU. This study involves collection and analysis of ultrasound exam results that are already being performed and documented as standard practice in our institution.

All pulmonary and critical care fellows who have attended the GNYHA ultrasound course during fellowship will be eligible for this study. Fellows also will attend pre-existing monthly lectures to discuss CCUS techniques and cases.

If a patient is to be evaluated in our study they should be newly admitted from the ER and the ultrasound assessment performed within 30 minutes of arrival to the medical intensive care unit. A fellow will document their initial indication for ultrasound on a standard assessment form followed by documentation of how much fluids the patient has received since admission. Based on the results of physical exam and ancillary testing the fellow will document pre-ultrasound diagnosis of shock and respiratory failure along with their initial assessment of whether the patient would respond to fluid bolus administration along with how much fluids the patient has gotten since arriving from the emergency room. This initial assessment will also be documented in the qpath database via the ultrasound machine. They will then document if they believe any diagnostic tests are indicated and the reason for ordering as well as any therapeutics indicated. They will then document their assessment of the diagnostic impact of the ultrasound exam to be performed.

A CCUS will then be performed on patients in shock or respiratory failure as is already protocol in our ICU. The ultrasound exam will be performed within 1 hour of arrival to the ICU. All images obtained will be saved to a password protected cloud database as is already our protocol. The ultrasound will require approximately 10 minutes and will not in hold up other tests or therapeutic interventions. The fellow will document the quality of images obtained and then pertinent findings on cardiac, lung, renal, vascular and abdominal exam.

Following performance of CCUS, the fellow will document post-ultrasound cause of shock, respiratory failure and volume responsiveness along with any other findings. They will then document if any diagnostic or therapeutic management changes are planned that differ from their pre ultrasound assessment and the reasons for the change in diagnostic or therapeutic plan.

An assessment of volume responsiveness using a CHEETAH non-invasive cardiac output hemodynamic monitor will then be performed directly after the ultrasound. This device is non-invasive and is already being used with frequency in the MICU, SICU and CCU of our institution to provide non-invasive assessment of whether a patient will respond to fluid challenge. The result of the test for volume responsiveness will be recorded on the standard assessment form.

All ultrasound exams will be submitted via the database for review by an attending expert clinician as is already standard practice in our training program. 72 hours following admission the ICU attending physician will be asked to document the final diagnosis and cause of shock or respiratory failure. The final diagnosis will be compared with the post-ultrasound diagnosis to measure the degree of variation.

The Phillips Sparq ultrasound is the machine most commonly used in our MICU. It has the ability to save images to a password protected cloud database and will thus be used in this study.

The study investigators will obtain all SAF's as well as the 'final' diagnosis from the attending physician at 72hours, and will enter this data into a database that will not contain any unique patient identifiers.

A waiver of informed consent will be requested in order to use the patients protected health information. This is appropriate since the research data will be de-identified and will not impact the patient's medical care.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted to the medical ICU.
* Clinical diagnosis of shock including systolic blood pressure less than 90 mmhg, patients requiring vasopressors or indication of organ hypoperfusion.
* Clinical diagnosis of respiratory failure including need for invasive or non-invasive mechanical ventilation, needing supplemental oxygen more than 50% face mask, clinical impression of respiratory failure with respiratory rate greater than 25.

Exclusion Criteria:

* Patients not in shock or respiratory failure based on the above criteria.
* Patients in shock but with obvious cause of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to our intensive care unit with shock and/or respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Diagnosis change | 5 minutes
  The proportion of times that clinical diagnosis changes following performance of a bedside ultrasound.
Management changes | 5 minutes
  The frequency and type of management changes that are made after performance of a critical care ultrasound.
Volume responsiveness agreement | 5 minutes
  The proportion of time that post-ultrasound assessment of volume responsiveness agrees with the volume responsiveness conclusion made by a cheetah monitor immediately after ultrasound is performed.

SECONDARY OUTCOMES:
Ultrasound diagnosis agreement with final diagnosis | 72 hours following admission to the ICU
  The proportion of the time that ultrasound diagnosis regarding etiology of shock and/or respiratory failure agrees with diagnosis 72 hours later in comparison to the pre-ultrasound clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kory, MD, Principal Investigator — Mount Sinai Beth Israel
Locations (1):
- Mount Sinai Beth Israel Medical Center, New York, New York, United States